CLINICAL TRIAL: NCT04058093
Title: VIVE Active: avaliação de um Programa de Treino Funcional Nos Cuidados de saúde primários - Estudo Quasi-experimental
Brief Title: Evaluation of a Functional Training Program in Primary Health Care
Acronym: VIVEactive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unidade de Saude da Ilha de Sao Miguel (Other)
Responsible Party: Principal Investigator, Sara B. Ponte, MD, General Practitioner, Unidade de Saude da Ilha de Sao Miguel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USISM_01_19
Record Dates: First submitted 2019-08-08; First posted 2019-08-15 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Sedentary Lifestyle
Keywords: Exercise; Physical activity; Nutrition; Counselling; Primary health care
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Training Program (Experimental): Functional training program (FTP) will last for 6 months and will include:
  1. Functional training sessions (each 45-minutes long, twice a week);
  2. Group nutrition counseling (each 90-minutes long, in three different moments throughout the intervention: week 1, 12 and 20).
  Interventions: Behavioral: Functional Training Program
- Waiting list control group (No Intervention): Participants will not participate in any specific intervention, but will receive the FTP after the experimental period (6 months).

INTERVENTIONS:
Behavioral: Functional Training Program — Functional training program (FTP) include:
  1. Functional training sessions will be oriented by graduates or masters in sport with the supervision of a sports medicine doctor;
  2. Group nutrition counseling, in the form of healthy cooking classes direct by nutritionists with the support of culinary students.
  Arms: Functional Training Program

SUMMARY:
Sedentarism is the fourth risk factor for worldwide mortality and morbility. Considering the high prevalence of sedentarism (57.0%) and obesity (30.5%) in Azores islands (Portugal), local primary health care (PHC) services should support the implementation of complementary interventions and the development of medical research in the area of active lifestyle promotion.

This study aims to evaluate the feasibility and effectiveness of a 6-months functional training program (FTP), which includes a group nutrition counseling, in sedentary users of Ponta Delgada Health Center (PDHC), compared to a waiting list control.

DETAILED DESCRIPTION:
This work will be a prospective, longitudinal, quasi-experimental study, with an experimental and a waiting list control group. Here, the investigators aim to test the feasibility and effectiveness of a 6-months functional training program in sedentary users of PDHC. The recruitment of participants will be held in PDHC by health professionals (e.g., family medicine doctors, nurses, nutritionists, psychologists, etc). Participants will be allocated into two groups (experimental and waiting list control groups). After signed informed consent and baseline measures, experimental group will conduct a 6-months functional training program (FTP), which comprises functional training sessions and group nutrition counseling. In every session, it will be evaluated the participants' adherence and theirs perceived enjoyment and exertion. The other outcomes (primary and secondary) will be analyzed through a face-to-face contact, in three different moments: baseline (T0), post-intervention (at month 6, T1) and 6-month follow-up (at month 12, T2). The control group will not participate in any specific intervention, but will receive the FTP after the experimental period. An intention-to-treat and per protocol analysis will be performed to analyze intervention effectiveness and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (<150 minutes of moderate-intensity PA per week or <75 minutes of vigorous-intensity PA) users of Health Center of Ponta Delgada.

Exclusion Criteria:

* Users with a medical contraindications to moderate-to-vigorous intensity physical activity, such as: unstable angina; deep vein thrombosis; recent thromboembolism or embolism; acute systemic infection or fever; atrioventricular block of 2nd grade or higher (without pacemaker); negative deflection of the ST segment deflection of the ST segment > 2 mm; severe neuro-musculoskeletal dysfunction; severe mitral or aortic insufficiency or stenosis without adequate treatment; decompensated heart failure; resting heart rate above 100 bpm; other decompensated metabolic disorders; pericarditis or acute myocarditis; uncontrolled arrhythmia; uncontrolled resting hypertension (SBP ≥ 180 or DBP ≥ 110); orthostatic hypotension with a fall in SBP> 20 mmHg or uncontrolled diabetes.
* Users with physical and/or mental disabilities or
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in hand grip strength | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Hand grip strength will be evaluated while the participant is in a sitting position with shoulders adducted and neutrally rotated, elbow flexed at 90°, forearm in neutral and wrist between 0 and 30° of extension. The test will be repeated 3 times with the dominant hand, and maximum reading will be taken.

SECONDARY OUTCOMES:
Adherence to the functional training program | Up to 6 months
  Proportion of adherence to the functional training program will be calculated by the average of adherence of each participant. The adherence of each participant will be quantified by the relationship between the sessions attended and the total number of sessions scheduled over the 6 months.
  Participants' satisfaction levels will be measured by 10-items questionnaire, on a five point Likert scale from 1 (displeased) to 5 (very satisfied).
Perceived enjoyment | Up to 6 months
  Perceived enjoyment of the functional training program will be measured biweekly by a scale rated from 1 (very unpleasant) to 5 (very enjoyable).
Perceived exertion | Up to 6 months
  Perception exertion the functional training program will be measured biweekly by the modified Borg scale. In this instrument, 11 items are evaluated, with a score of 0 to 10 points, where 0 equals the minimum effort and 10 the maximum that they can perform.
Participants' satisfaction | T1, Post-intervention (at month 6)
  Participant's satisfaction levels will be measured by 10-items questionnaire, on a five point Likert scale from 1 (displeased) to 5 (very satisfied).
Change in body mass index | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Weight (kilograms) and height (meters) will be combined to report BMI in kg/m^2.
Change in waist circumference | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Waist circumference in centimeters.
Change in body fat | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Measured by bioelectrical impedance analysis.
Change in body lean mass | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Measured by bioelectrical impedance analysis.
Change in systolic and diastolic blood pressure | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Resting systolic and diastolic blood pressure.
Change in fast blood glycemia | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Fast blood glycemia (mg/dL).
Change in HbA1c | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  HbA1c (%) reflects the average plasma glucose over the previous 8 to 12 weeks.
Change in blood lipid profile | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides.
Change in chronic pain | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Brief Pain Inventory (BPI) will assess the average pain at rest, using a numerical (0-10) rating scale on the BPI Short Form. A higher score indicates worse pain (10 is "worst pain imaginable") and zero indicates 'no pain at all'.
Change in medication dependence | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Number of pills ingested per day (includes antihypertensives, oral antidiabetics, insulin (injected units), analgesics, anti-inflammatory drugs, psychotropic drugs and antidyslipidemic).
Change in nicotine dependence | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Fagerström Test for Nicotine Dependence (FTND) will be applied only in smokers participants.
  FTND is a 6-item self-report measure of nicotine dependence derived from the Fagerström Tolerance Questionnaire, which comprises yes/no options (scored from 0 to 1) and multiple-choice items (scored from 0 to 3). The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
Change in health-related quality of life | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  The health-related quality of life questionaire EQ-5D-5L is a standardised self-report measure of health status developed by the EuroQol Group. It consists of the descriptive system and the EQ Visual Analogue scale. The descriptive system comprises 5 dimensions, namely mobility, self care, usual activities, pain/discomfort, anxiety/depression.
Change in perceived stress | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Perceived Stress Scale (PSS 10), validated for portuguese population, is a self-report scale with 10 items on daily hassles and the current feeling of being able to handle problems that need to be addressed. It is a five-point Likert scale ranging from 0 (never) to 4 (very often). This questionnaire is widely used to measure perceived stress and has adequate internal and test-retest reliability.
Change in psychological distress | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Depression, anxiety stress scale-21 (DASS-21) consists of three 7-item subscales: depression, anxiety, and stress. Participants indicate how much each of 21 items applies to them over the past week on a scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). This scale has good psychometric properties in both clinical and non-clinical samples. Also, this scale reliably distinguishes between symptoms of anxiety (panic/worry), stress (tension/agitation) and depression (low mood/anhedonia), which are highly comorbid.
Change in mental well-being | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  Warwick-Edinburgh Mental Well-being Scale (WEMWBS) is a 14-item scale, validated and self-report instrument used to assess mental wellbeing in general population. Possible scores range from range from 14-70, with higher scores indicating higher mental well-being.
Changes in eating habits | T0, baseline; T1, post-intervention (at month 6); and T2, 6-month follow-up (at month 12)
  PREDIMED (PREvención con DIeta MEDiterránea) is a questionnaire to assess the adherence to the Mediterranean diet, 0 being the minimum total score and 14 the maximum total score. Higher values represent a higher adherence to the Mediterranean diet.

CONTACTS AND LOCATIONS:
Overall Officials: Sara B. Ponte, MD, Principal Investigator — Unidade de Saúde da Ilha de São Miguel
Locations (1):
- Centro de Saúde de Ponta Delgada (Unidade de Saúde da Ilha de São Miguel), Ponta Delgada, Azores, Portugal